CLINICAL TRIAL: NCT06735898
Title: Evaluation of the Efficacy of Permanent Course Combined Therapy With CYTOFLAVIN® Intravenous Solution and CYTOFLAVIN® Tablets, at 2-3 Stages of Rehabilitation of Patients With Post Intensive Care Syndrome
Brief Title: Evaluation of the Efficacy of Permanent Course Combined Therapy With CYTOFLAVIN® Intravenous Solution and CYTOFLAVIN Tablets, at 2-3 Stages of Rehabilitation of Patients With Post Intensive Care Syndrome
Status: Recruiting | Type: Observational
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Other Study IDs: PR-C_2
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Ischemic Stroke
Keywords: Post Intensive Care Unit Syndrome; Ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Basic therapy + Cytoflavin® intravenous solution in the volume of 20 ml per day IV drip in dilution on 100-200 ml of 5-10% dextrose solution or 0.9% sodium chloride solution during 10 days, transition to Cytoflavin® tablets from the next day after the end of intravenous administration during the next 75 days according to the instructions for medical use
- Group 2: Basic therapy, according to clinical guidelines (clinical practice established within the center) for the treatment of patients in stages 2-3 of rehabilitation.

SUMMARY:
Post intensive care syndrome (PIC syndrome) is an important problem in modern intensive care strategy. Understanding the mechanisms of PIC syndrome helps prevent it in patients with respiratory, neuromuscular transmission, and cognitive impairments that require prolonged support of vital functions. Significant role in the formation and severity of PIC syndrome is played by the severity of the systemic inflammatory response, which is an individual reaction of the body, and this determines the degree of neurological and psychological deficits. Chronic diseases such as diabetes mellitus, especially in the context of metabolic syndrome, worsen the course of PIC syndrome and delays recovery. Early initiation of rehabilitation measures in the intensive care unit and subsequent expansion of the individual rehabilitation program contributes to the rapid and successful recovery of not only vital functions, but also cognitive, motor and emotional disorders. This shortens the hospital stay of patient and improves their quality of life after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years of age and older;
* Stay in the ITU and (or) intensive care unit for at least 3 days;
* Diagnosed "post intensive care" syndrome (PIC syndrome) with moderate-to-severe severity >3<6 points
* Diagnosed modalities "critical illness polyneuropathy, respiratory neuropathy, dysphagia" of the domain "Neuromuscular complications" of PIC syndrome at 2-3 stages of the rehabilitation route at any value of PICS severity index
* Diagnosed modalities "decreased gravitational gradient, decreased exercise tolerance" in the domain "Vegetative-metabolic complications" at 2-3 stages of the rehabilitation route at any value of PICS severity index

Exclusion Criteria:

* Premorbid level of vital activity when assessed on the rehabilitation routing scale 4-5 points;
* Hematocrit ≤30%;
* Hemoglobin level ≤80 g/L;
* Acute cardiac failure;
* Acute respiratory failure;
* Acute renal failure;
* Acute liver cell failure;
* Use of drugs from "metabolic agents" pharmacotherapeutic group at the time of inclusion in the study
* Life expectancy of 6 months or less or presence of incurable diseases in decompensation stage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The observational program will include adult patients of both sexes with signs of PIC syndrome after a stay in Anesthesiology, reanimation and intensive treatment department due to acute cerebral insufficiency for at least 72 hours, hospitalized for stage 2-3 rehabilitation in a rehabilitation center between 14 and 60 days after the onset of the disease.
  The group of patients who received Cytoflavin at stage 1 during the RehabIT program will be "automatically" allocated to the Basic Therapy + Cytoflavin group
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Dynamics of rehabilitation routing status score | day 12, day 30, day 60, day 90
  Dynamics of rehabilitation routing status score from the start of the study (Visit 1) to Visit 3, Visit 4, Visit 5 and Visit 6 measured in both groups
Dynamics of Barthel status score | day 12, day 30, day 60, day 90
  Dynamics of Barthel status score from the start of the study (Visit 1) to Visit 3, Visit 4, Visit 5 and Visit 6 measured in both groups
Dynamics of EQ5 status score | day 12, day 30, day 60, day 90
  Dynamics of EQ5 status score from the start of the study (Visit 1) to Visit 3, Visit 4, Visit 5 and Visit 6 measured in both groups

SECONDARY OUTCOMES:
Dynamics of somatic status | day 12, day 30, day 60, day 90
  Dynamics of somatic status from the start of the study (Visit 1) to Visit 3, Visit 4, Visit 5 and Visit 6 measured in both groups
Dynamics of rehabilitation status | day 12, day 30, day 60, day 90
  Dynamics of rehabilitation status from the start of the study (Visit 1) to Visit 3, Visit 4, Visit 5 and Visit 6 measured in both groups

OTHER OUTCOMES:
Identification during the event related monitoring of responders and non-responders | day 12, day 30, day 60, day 90
  Identification during the event related monitoring of responders and non-responders for the use of cytoflavin for adjunctive drug modulation in PIT syndrome rehabilitation

CONTACTS AND LOCATIONS:
Locations (1):
- Brain Institute Clinic, Yekaterinburg, Sverdlovsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: No